CLINICAL TRIAL: NCT02335333
Title: Clinical Utility of Biomarkers of Aging as Predictors of Kidney Graft Function in Extended Criteria Organ Recipients
Brief Title: Biomarkers of Aging as Predictors of Kidney Transplant Function
Status: Completed | Type: Observational
Sponsor: Sapere Bio (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: HSDX-1501
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Delayed Graft Function; Other Complications of Kidney Transplant
Keywords: Delayed Graft Function; Slow Graft Function; Renal Transplant; Extended Criteria Donor; Biomarker of Aging; Kidney Transplant
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — T lymphocytes, plasma and white blood cells isolated from peripheral blood sample will be stored.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No treatment

SUMMARY:
The primary purpose of this study is to measure the correlation between baseline expression of aging biomarkers, SenesceTest in blood of organ donor and renal graft function. This pilot study will study patients who are undergoing renal transplantation with organs from extended criteria donors, standard criteria donors or donation after cardiac death and compare ability of SenesceTest to predict renal graft function immediately after the transplant and at 1 year followup.

DETAILED DESCRIPTION:
Presently, donated organs are ranked amongst each other based on a formula for Kidney Donor Patient Index (KDPI; a variation of Donor Risk index) 8 which includes donor demographics and clinical history but no molecular markers of kidney function other than serum creatinine. Using KDPI assessment, nearly all ECD kidneys fall into the high-risk category. And while ECD kidneys are associated with higher risk of graft failure, studies note a wide variability in ECD organ quality and the associated graft survival (half-life graft survival 4.5-7.9 years), suggesting that current models of assessing organ quality are inadequate. Furthermore, prior to even being assigned a KDPI, over 37% of all kidneys and over 50% of ECD kidneys are discarded based on biopsy findings. However, recent studies called into question the reliance on procurement kidney biopsy reports in making acceptance decisions by demonstrating significant overlap in the biopsy findings between discarded and transplanted kidneys. The use of ECD kidneys is becoming more widespread and, according to a recent report, 70% adults >65yo and 50% adults between 50 and 64 yo are willing to accept an ECD kidney. Therefore, new methodology for assessment of graft viability would increase transplantation rates particularly for organs from older or expanded criteria donors, shorten patient's time on wait list (currently 45 months average 50) and improve their outcomes by taking them off dialysis sooner.

Here, we propose a new approach-using molecular age markers (collectively referred to as SenesceTest) to predict kidney graft function.

ELIGIBILITY:
Inclusion Criteria:

* Donor > 35 years of age

Exclusion Criteria:

* Recipient is HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal Transplant Recipients at UNC Hospitals who received a single organ from a deceased donor (ECD, DCD, or SCD).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Slow graft function (SGF; decline in serum creatinine >20% within 24h after transplant, no dialysis) | 24h
Delayed graft function (DGF; need for dialysis during first week after transplant) | 1 week

SECONDARY OUTCOMES:
Long-term graft function measured by change in serum creatinine (delta1-12eGFR) | 12 months
Long-term graft function measured by change in serum creatinine (delta1-6eGFR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Gerber, MD, Principal Investigator — University of North Carolina- Department of Surgery
Locations (2):
- United States (2):
  - UNC Hospitals, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Abdominal Organ Transplant Program, Winston-Salem, North Carolina